CLINICAL TRIAL: NCT00825591
Title: Identification and Treatment of Biological Clock Dysfunction in Optic Nerve Hypoplasia
Brief Title: Biological Clock Dysfunction in Optic Nerve Hypoplasia
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Children's Hospital Los Angeles (Other)
Responsible Party: Esther Nakamura-Reyes, Childrens Hospital of Los Angeles
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: 0804003699; TRSH-SAR
Record Dates: First submitted 2008-10-13; First posted 2009-01-21 (Estimated); Last update posted 2020-09-25 (Actual); Status verified 2020-09

CONDITIONS: Biological Clock Dysfunction; Optic Nerve Hypoplasia
Keywords: optic nerve hypoplasia; septo-optic dysplasia; melatonin; circadian rhythm
MeSH Terms: conditions — Optic Nerve Hypoplasia; Septo-Optic Dysplasia | interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Individuals with abnormal rhythmicity will be treated with melatonin to assess if sleep patterns are improved.
  Interventions: Dietary Supplement: Melatonin
- 2 (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo Comparator

INTERVENTIONS:
Dietary Supplement: Melatonin — Oral administration before bed. We will test two doses (0.5 or 3.0 mg/m2. 6 week duration.)
  Arms: 1
Dietary Supplement: Placebo Comparator — Oral administration before bed. 6 week duration.
  Arms: 2

SUMMARY:
Background: Optic Nerve Hypoplasia (ONH) is a leading cause of blindness in children. For unclear reasons, the incidence of ONH is increasing, with ONH affecting about 1 in 10,000 live-born infants. In addition to visual deficits, ONH is associated with varying degrees of hypopituitarism, developmental delay, brain malformations and obesity. Although genetic mutations have been rarely observed to result in ONH, the causes of ONH are largely not known. In limited anatomical observations, the suprachiasmatic nuclei (SCN) located in the anterior hypothalamus, which generate circadian rhythms, have been observed to be abnormal in children with ONH. Thus, children with ONH may have biological clock dysfunction.

In collaborative studies with Dr. Mark Borchert of Childrens Hospital Los Angeles (CHLA), we have recently discovered that one-half of children with ONH have grossly abnormal sleep-wake patterns, as assessed by actigraphy. Although not known for children with ONH, abnormal sleep-wake patterns have been observed to be associated with neurocognitive impairment and obesity. We also observe that nocturnal melatonin administration can improve abnormal sleep-wake cycles in these children, raising the possibility that it will be possible to treat abnormal rhythmicity in children with ONH.

DETAILED DESCRIPTION:
Objectives and Hypotheses. Our objectives are to define the scope and problems related to biological clock disorders in children with ONH and to develop effective treatments for this condition. Based on our observations, we hypothesize: (1) Daily rest-activity patterns and sleep will be abnormal in up to 50% of children with ONH. (2) It is possible to identify risk factors for abnormal circadian system function and sleep problems in ONH. (3) Nocturnal melatonin administration will improve abnormal sleep and activity patterns in children with ONH.

Design: These studies will involve collaborative efforts between Yale University and Dr. Mark Borchert of Childrens Hospital Los Angeles, who follows the largest population of children with ONH in the world. We will study children ages 2-10 years with documented ONH using standard criteria. Based on these criteria, we have more than 100 eligible patients.

To test our hypotheses, we will: (1) examine expressed rhythmicity in children with ONH. These studies will use actigraphy, sleep questionnaires, and assessment of melatonin secretory profiles. (2) We will correlate hypothalamic anatomical abnormalities and the degree endocrine dysfunction with sleep and expressed rhythmicity. (3) We will test if short-term administration of melatonin improves sleep-wake patterns in children with abnormally-expressed rhythmicity.

Potential Impact: Our preliminary data raise the possibility that children with ONH will have circadian system dysfunction resulting in abnormal rhythmicity and sleep. However, to date there have been no formal attempts to identify children with ONH who are at risk for such problems, nor have there been efforts aimed at developing potential treatments. The proposed prospective clinical study will represent an important attempt to identify a group of children with circadian system dysfunction.

At the completion of this study, we anticipate having determined risk factors for circadian system dysfunction in children with ONH. Insights gained from these studies should lead to the development of new approaches for treating circadian clock lesions in ONH, with the hope of improving the well-being of circadian system function in the boys and girls with this condition.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of ONH (Diagnosis will be confirmed by ocular fundus photography.Disc-macula distance 0.35 or below. In eyes without ONH, the DD/DM ratio is greater than 0.3581.)
* Ages 2-10 years
* Ability to ambulate independently
* Under care of endocrinologist if on pituitary hormone replacement therapy.

Exclusion Criteria:

* Non-ambulatory
* Active malignancy
* Cardio-respiratory disorder

Ages: 2 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2008-10 (Actual); Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Assessment of rest-activity patterns | two years

CONTACTS AND LOCATIONS:
Overall Officials: Casandra Fink, Study Director — Children's Hospital Los Angeles
Locations (1):
- Children's Hospital of Los Angeles, Los Angeles, California, United States